CLINICAL TRIAL: NCT00961844
Title: Phase I/II Trial for Vaccine Therapy With Dendritic Cells - Transfected With hTERT-, Survivin- and Tumor Cell Derived mRNA + ex Vivo T Cell Expansion and Reinfusion in Patients With Metastatic Malignant Melanoma
Brief Title: Trial for Vaccine Therapy With Dendritic Cells in Patients With Metastatic Malignant Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Logistical problems
Sponsor: Steinar Aamdal (Other)
Responsible Party: Sponsor-Investigator, Steinar Aamdal, MD, PhD, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC-004; 2008-006253-41 (EudraCT Number)
Record Dates: First submitted 2009-08-12; First posted 2009-08-19 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Metastatic Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Survivin; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DC vaccine + Temozolomide (Experimental): Dendritic cell loaded with h-TERT mRNA, survivin mRNA and autologous tumor cell mRNA, lymphodepletion treatment and T cell expansion and reinfusion.
  Interventions: Biological: Dendritic cells - transfected with hTERT-, survivin- and tumor cell derived mRNA + ex vivo T cell expansion and reinfusion; Drug: Temozolomide

INTERVENTIONS:
Biological: Dendritic cells - transfected with hTERT-, survivin- and tumor cell derived mRNA + ex vivo T cell expansion and reinfusion
Drug: Temozolomide

SUMMARY:
In this trial the investigators want to combine chemotherapy with immunotherapy by giving the patients Temozolomide, before vaccination. The investigators have also included hTERT and survivin mRNA in the vaccine. Finally, the investigators want to introduce ex vivo T cell expansion after lymphodepletion for the patients who show an immune response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified malignant melanoma with measurable (according to RECIST), unresectable metastases (Stage III or Stage IV M1a-c as defined by criteria of the AJCC Cancer Staging Manual, 6 th. Edition 2002). Patients with a melanoma of an unknown primary site are eligible.
* Preferably accessible tumor tissue with enough volume and quality for vaccine production (extraction of tumor mRNA)
* Must be at least 18 years of age
* Must be ambulatory with a ECOG performance status 0 or 1
* Life expectancy ≥ 6 months
* Negative MRI of the brain
* Must have lab values as the following:

  * ANC ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hb ≥ 9 g/dL (≥ 5.6 mmol/L)
  * Creatinine ≤ 140 μmol/L (1.6 mg/dL); if borderline, the creatinine clearance ≥ 40 mL/min
  * Bilirubin < 20% above the upper limit of normal
  * ASAT and ALAT ≤ 2.5 the upper limit of normal
  * Albumin ≥ 2.5 g/L
* If the patient is female, she must practice adequate contraception during the study treatment
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* The patient suffers from an ocular- or mucous membrane melanoma
* History of prior malignancy other than melanoma, except for curatively treated basal cell or squamous cell carcinoma of the skin and cervix cancer stage 1B or effectively treated malignancy that has been in remission for over 5 years and is highly likely to have been cured.
* Active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune systems. PI shall make the final determination regarding appropriateness of enrollment
* Autoimmune disease currently being treated with systemic steroids Version no. 3, 18 June 2009 Page 17 of 50
* Adverse reactions to vaccines such as anaphylaxis or other serious reactions
* History of immunodeficiency or autoimmune disease such as rheumatoid arthritis, systemic lupus erythematosus, scleroderma, polymyositis-dermatomyositis, juvenile onset insulin dependent diabetes, or a vasculitic syndrome
* Positive for HIV, Hepatitis B and C and Syphilis (treponema pallidum)
* Pregnancy or lactation
* If the patient has received any prior anti-cancer treatment, including radiotherapy, chemotherapy immunotherapy and/or immunomodulating agents, this must have been stopped at least 4 weeks before first study treatment administration.
* Chemotherapy, glucocorticosteroids or other potentially immune-suppressive therapy that has been administered within 4 weeks prior to vaccination
* No treatment with dacarbazine or temozolomide at any time prior to study entry
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity of vaccination with DC transfected h-TERT mRNA, survivin mRNA and tumor cell mRNA, lymphodepletion treatment and T cell expansion and reinfusion in patients with metastatic malignant melanoma.

SECONDARY OUTCOMES:
Evaluation of immunological responses, time to disease progression and survival time. | 5 years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Aamdal, M.D PhD Prof, Principal Investigator — Oslo University Hospital - Norwegian Radium Hospital
Locations (1):
- The Norwegian Radium Hospital, Department of Clinical Cancer Research, Oslo, Montebello, Norway